CLINICAL TRIAL: NCT02352766
Title: Role of NGS-based ThyroSeq Panel in Cancer Diagnosis in Thyroid Nodules
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Duke University (Other); Johns Hopkins University (Other); Ohio State University (Other); University of Cincinnati (Other); University of Colorado, Denver (Other); University of Pennsylvania (Other); University of Wisconsin, Madison (Other); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Yuri Nikiforov, Professor of Pathology; Vice Chair for Molecular Pathology, University of Pittsburgh
Other Study IDs: PRO14040164; PITT 9006477 (Other Grant/Funding Number: University of Pittsburgh)
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Thyroid Nodule
Keywords: Thyroid cancer; Thyroid nodules; Palpable nodules; FNA
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Routine FNA for thyroid nodules: Patients that undergo a clinically diagnostic thyroid FNA will be asked by their clinician, who is a study co-investigator, if they are interested in participating in the research study. A small part of FNA material will be collected for molecular analysis.

SUMMARY:
Recently, targeted next generation sequencing (NGS) platforms have been introduced that allow inexpensive testing for hundreds of mutational hotspots at the same time. A number of additional mutational markers in thyroid cancer have been identified. Highly promising markers associated with tumor prognosis have also been found. This multi-institutional study aims to validate the diagnostic use of mutational markers in thyroid nodules with indeterminate cytology.

The proposed hypothesis is that a broad NGS-based genotyping of thyroid nodules using a large panel of mutational markers applied to thyroid FNA samples can provide an accurate cancer risk stratification in thyroid nodules.

The performance of the panel will be tested in a multi-institutional double-blind prospective study of FNA samples from thyroid nodules with indeterminate cytology and available surgical outcome

DETAILED DESCRIPTION:
Thyroid cancer is the fifth most common cancer type in women and the fastest growing cancer diagnosis in the U.S. In 2013, an estimated 60,000 new cases were diagnosed. However, thyroid nodules are much more common, particularly in woman and with increased age. The prevalence of palpable nodules in population-based studies is 3-4% and the prevalence of non-palpable nodules incidentally identified on imaging approaches 40-50% after the age of 60. Thyroid cancer is the primary clinical concern in patient with thyroid nodules, although only small proportion (~5%) of thyroid nodules is malignant . The diagnosis of thyroid cancer relies on cervical ultrasound and fine needle aspiration (FNA) biopsy with cytologic examination. FNA cytology provides a definitive diagnosis of benign or malignant thyroid disease in most cases, although in approximately 30% of nodules, FNA cytology cannot reliably rule out cancer and such cases are reported as indeterminate for malignancy. Because of the lack of a definitive diagnosis, most patients with indeterminate cytology undergo diagnostic surgery to establish histopathologic diagnosis. However, only 20-30% of such surgically resected thyroid nodules will prove to be malignant. It has been estimated that ~150,000 thyroid surgeries are performed in the U.S. for benign nodules due to inability to rule out cancer without surgery. Additionally, an indeterminate preoperative diagnosis does not always lead to the optimal initial surgical intervention for patients who have thyroid cancer, as many of them undergo a two-step surgery, i.e. thyroid lobectomy followed by completion total thyroidectomy. Both unnecessary and two-step surgeries can be avoided with a more accurate preoperative diagnosis of cancer in thyroid nodules.

For patients who have signed an informed consent, the physician investigator will then perform a research needle wash. The syringe will be rinsed with a buffer solution to gather left over cells for the research sample. This FNA material will be collected for potential molecular testing into a collection tube that is stored at -20C.

The first five samples acquired will be processed irrespective of cytologic diagnosis to evaluate the collection technique.

Those samples that have indeterminate cytologic diagnosis (Bethesda III, VI, or V) and surgical outcome are submitted for molecular testing. (Sample will be given a code that de-identifies the sample before it is sent to the testing laboratory. The lab that will analyze specimens is a CLIA certified Pitt lab.)

Molecular analysis is performed at the Pitt lab without knowing surgical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients that undergo a clinically diagnostic thyroid FNA

Exclusion Criteria:

* Children
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that undergo a routine diagnostic thyroid FNA that consent in participating in the research study whose samples have indeterminate cytologic diagnosis (Bethesda III, VI, or V) and surgical outcome are submitted for molecular testing. (Sample will be given a code that de-identifies the sample before it is sent to the testing laboratory. The lab that will analyze specimens is a CLIA certified Pitt lab.)
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2015-01; Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Primary outcomes | April 2016
  The primary outcome measured in this study is the performance (sensitivity, specificity, NPV, PPV) of the Thyroseq Panel in diagnosing cancer in thyroid nodules with Bethesda III, VI and V cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Nikiforov, PhD, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States